CLINICAL TRIAL: NCT05348135
Title: Synergistic Effect of Functional Strength Training and Cognitive Intervention on Motor and Cognitive Functions in Children With Cerebral Palsy
Brief Title: Combined Cognitive and Functional Strength Training in Children With cp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fahmy Hassan Al Nemr, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/003398
Record Dates: First submitted 2022-03-12; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Functional strength training (Active Comparator)
  Interventions: Other: functional strength training
- Cognitive training (Active Comparator)
  Interventions: Other: cognitive training
- Combined treatment (Active Comparator)
  Interventions: Other: functional strength training; Other: cognitive training
- Conventional physical therapy (Placebo Comparator)
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: functional strength training — children in this group received FST. Each training session started with 10 minutes dynamic warm-up period and ended with 5 minutes cool down in the form of muscle stretching and aerobics. The warm up was followed by gait training in addition to 4 functional lower limb exercises; sit to stand exercise, forward/ lateral step-up exercise, half knee rise exercise, and bridging exercise.
  Arms: Combined treatment; Functional strength training
Other: cognitive training — Children in this group received cognitive training by RehaCom cognitive rehabilitation software. Training was applied for four cognitive domains of function; attention / concentration, figural memory, reaction behavior and logical reasoning.
  Arms: Cognitive training; Combined treatment
Other: conventional physical therapy — including reinforcement of normal motor development, reflex inhibiting patterns, balance exercises, stretching exercises and gait training
  Arms: Conventional physical therapy

SUMMARY:
Cerebral palsy is primarily a disorder of movement and posture however; it often involves disorder of different aspects of cognitive function.

DETAILED DESCRIPTION:
This study evaluated the effect of FST and cognitive intervention and their combined effect on motor and cognitive functions in children with spastic diplegia. A convenient sample of spastic diplegic CP children, with their age ranging from 8 to 12 years were assigned randomly into four treatment groups

ELIGIBILITY:
Inclusion Criteria:

* chronological age ranged from 8 to 12 years,
* spasticity grade in affected lower limbs ranged between 1 + and 2 according to MAS
* can follow instructions given to them,
* their intelligence level ranged from 65 to 80 according to Stanford Binet intelligence scale, - -- their motor function ranged between Level II & III according to Gross Motor Functional Classification System Expanded and Revised (GMFCS E&R).

Exclusion Criteria:

* children who had visual or auditory problems
* children who took any medicine affecting alertness
* fixed deformities in the joints of upper & lower limbs
* any orthopedic surgery in lower limbs within 6 months before study
* epileptic children.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
change in GMFM-88 measures | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  criterion-referenced scale that measure gross motor function in children with CP.
change in attention / concentration measures | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  * Computer based RehaCom software used to assess attention / concentration cognitive domain of function. It is clinically proven and evidence-based software.
  * minimum reaction time ( in seconds) of attention / concentration program was assessed
change in figural memory measures | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  * Computer based RehaCom software used to assess figural memory cognitive domain of function.It is clinically proven and evidence-based software.
  * minimum reaction time ( in seconds) of figural memory program was assessed
change in reaction behavior measures | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  Computer based RehaCom software used to assess reaction behavior cognitive domain of function. It is clinically proven and evidence-based software.
  - minimum reaction time ( in seconds) of reaction behavior program was assessed
change in logical reasoning measures | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  Computer based RehaCom software used to assess logical reasoning cognitive domain of function. It is clinically proven and evidence-based software.
  - minimum reaction time ( in seconds) of logical reasoning program was assessed

SECONDARY OUTCOMES:
change in Five times sit to stand test (FTSST) measure | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  measure the time spent for completing five sequential sit to stand to sit cycles. It is a reliable and valid measure of functional muscle strength and balance in CP children.
change in Timed up and go test (TUG)measure | The assessment was performed 3 times; at baseline, 6 months (post-treatment) and at 6 months follow up
  A reliable and valid test used for assessing dynamic balance and functional mobility in the children.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No